CLINICAL TRIAL: NCT04598542
Title: Open-Label, Parallel-Arm Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Corticosteroid Intra Articular Injection Given 7 Days Before or 7 Days After Lorecivivint Intra-articular Injection Into the Knee of Healthy Volunteers
Brief Title: Drug-Drug Interaction Study of Lorecivivint and Triamcinolone Acetonide in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SM04690-OA-16
Record Dates: First submitted 2020-10-06; First posted 2020-10-22 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Drug-Drug Interaction
Keywords: lorecivivint; triamcinolone acetonide
MeSH Terms: interventions — lorecivivint; Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TA injection followed by LOR injection (Experimental): IA injection of TA into the right knee, followed by IA injection of LOR into the same knee 7 days later.
  Interventions: Drug: Lorecivivint (LOR); Drug: Triamcinolone acetonide (TA)
- LOR injection followed by TA injection (Experimental): IA injection of LOR into the right knee, followed by IA injection of TA into the same knee 7 days later.
  Interventions: Drug: Lorecivivint (LOR); Drug: Triamcinolone acetonide (TA)

INTERVENTIONS:
Drug: Lorecivivint (LOR) — 0.07 mg
  Other Names: SM04690
Drug: Triamcinolone acetonide (TA) — 40 mg

SUMMARY:
This study will be an open-label, parallel-arm study to determine if a prior intra-articular (IA) injection of lorecivivint (LOR) affects the safety, tolerability, and/or pharmacokinetics (PK) of a subsequent IA injection of the corticosteroid triamcinolone acetonide (TA) into the same knee, and to determine if a prior IA injection of TA affects the safety or tolerability of a subsequent IA injection of LOR into the same knee.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males and females between 18 and 55 years of age, inclusive, in general good health
2. Body mass index (BMI) ≥ 18.5 and ≤ 32.0 kg/m2 at Screening
3. Negative drug test for amphetamine, cocaine, methadone, opiates, phencyclidine (PCP), barbiturates, benzodiazepines, tricyclic antidepressants, and marijuana

Key Exclusion Criteria:

1. Pregnant women, breastfeeding women, and women who are not post-menopausal (defined as 12 months with no menses without an alternative medical cause) or permanently surgically sterile (includes hysterectomy, bilateral salpingectomy, and bilateral oophorectomy) who have a positive or indeterminate pregnancy test result at the Screening Visit or Day -1
2. Women who are not post-menopausal or permanently surgically sterile who are sexually active, and who are not willing to use birth control during the study period
3. Men who are sexually active and of reproductive potential, who have partners who are capable of becoming pregnant, and who are not willing to use birth control during the study period
4. Any chronic medical condition that requires medication
5. Any history of IA injection, surgery (e.g., arthroscopy), infection, major orthopedic injury, or inflammatory rheumatic diseases (e.g., rheumatoid arthritis, gout, pseudogout) of either knee
6. Any contraindications for an IA injection in the right knee in the opinion of the Investigator
7. Previous treatment with lorecivivint (LOR)
8. Treatment with any glucocorticoids (oral, intravenous, intramuscular, IA, topical, or inhaled) within 12 weeks before Day 1
9. Consumption of grapefruit, grapefruit juice, Seville oranges, or vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, brussels sprouts) within 10 days before Day 1
10. Known hypersensitivity to triamcinolone acetonide (TA)
11. Significant blood loss (> 500 mL) or donation of blood within 30 days of screening
12. Regular use of nicotine-containing products, including, but not limited to, cigarettes, e-cigarettes, or nicotine gum or patches
13. Any condition, that, in the opinion of the Investigator, constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation
14. Estimated glomerular filtration rate (eGFR) of < 60 mL/min/1.73 m2, calculated using the Modification of Diet in Renal Disease (MDRD) equation at the Screening Visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Cmax of LOR | 0, 0.25, 0.5, 1, 2, 4, 6, 8 hours after administration
AUC 0-last of LOR | 0, 0.25, 0.5, 1, 2, 4, 6, 8 hours after administration
Plasma concentration profiles of LOR | 0, 0.25, 0.5, 1, 2, 4, 6, 8 hours after administration
Cmax of TA | 0, 1, 2, 4, 6, 8, 10, 12, 24, 48, 96 hours after administration
AUC 0-last of TA | 0, 1, 2, 4, 6, 8, 10, 12, 24, 48, 96 hours after administration
Plasma concentration profiles of TA | 0, 1, 2, 4, 6, 8, 10, 12, 24, 48, 96 hours after administration

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Yazici, M.D., Study Director — Biosplice Therapeutics, Inc.
Locations (1):
- Research Site, Miami, Florida, United States

REFERENCES:
- [Derived] Fineman MS, McAlindon TE, Lattermann C, Swearingen CJ, Kennedy S, Lopez VA, Simsek I, Tambiah JRS, Yazici Y. Safety, Tolerability, and Pharmacokinetics of Same-Knee Intra-Articular Injection of Corticosteroid and Lorecivivint Within 7 Days: An Open-Label, Randomized, Parallel-Arm Study. Rheumatol Ther. 2023 Dec;10(6):1741-1752. doi: 10.1007/s40744-023-00604-7. Epub 2023 Oct 30. PMID 37902943